CLINICAL TRIAL: NCT01429701
Title: Unicentric Comparing Effectiveness of Polymyxin B Sulphate + Prednisolone + Benzocaine + Clioquinol to Betamethasone + Gentamicin + Tolnaftate + Clioquinol in Acute and Sub-acute Dermatitis Eczematous
Brief Title: Effectiveness of Polymyxin B Sulphate + Prednisolone + Benzocaine + Clioquinol in Acute and Sub-acute Dermatitis Eczematous
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREEMS0711
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2013-03

CONDITIONS: Eczema
Keywords: Dermatitis; Dermatitis, Atopic
MeSH Terms: conditions — Eczema; Dermatitis; Dermatitis, Atopic | interventions — Polymyxin B; Prednisolone; Benzocaine; Clioquinol; Betamethasone; Gentamicins; Tolnaftate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test association cream (Experimental): polymyxin B sulphate + prednisolone + benzocaine + clioquinol
  Interventions: Drug: polymyxin B sulphate + prednisolone + benzocaine + clioquinol
- Comparative association cream (Active Comparator): betamethasone + gentamicin + tolnaftato + clioquinol
  Interventions: Drug: betamethasone + gentamicin + tolnaftato + cleoquinol

INTERVENTIONS:
Drug: polymyxin B sulphate + prednisolone + benzocaine + clioquinol — applied 3 times / day at lesion
  Arms: Test association cream
Drug: betamethasone + gentamicin + tolnaftato + cleoquinol — applied 3 times / day at lesion
  Arms: Comparative association cream

SUMMARY:
Dermatitis eczematous is a recurrent pruritic skin disorder which has a significant morbidity and impaired quality of life due specially pruritus and physical visible skin lesions. The purpose of this trial is evaluate the effectiveness of two different topic associations of drugs.

DETAILED DESCRIPTION:
Study design:

* Experiment duration: 22 days
* 2 visits (days 0,7,15 and 22)
* Reducing eczema area and severity index evaluation
* Adverse events evaluation
* Double blinded, non-inferiority, prospective parallel-group, intend to treat trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Patients with acute or subacute dermatitis with a minimum of 3 symptoms.

Exclusion Criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation
3. Use of anti-inflammatory or immunosuppressive drugs (last 30 days prior to the study).
4. Sunlight over exposure in the last 15 days.
5. Any pathology or past medical condition that can interfere with this protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Reduction / improvement of signs and symptoms | DAY 22
  The reduction of signs and symptoms will be evaluated by OSAAD index.

SECONDARY OUTCOMES:
Adverse Events Evaluation | DAY 22
  Adverse events will be collected and followed in order to evaluate safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Flávia Addór, MD., Principal Investigator — Medicin Instituto da Pele